CLINICAL TRIAL: NCT06364943
Title: Application of Tear Ferning Test for Clinical Dry Eye Diagnosis
Brief Title: Tear Ferning Test for Dry Eye Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, David Pei-Cheng Lin, Chung Shan Medical University, Chung Shan Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202400020B0
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye diagnosis; Tear ferning
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry eye patients (No Intervention): Collect clinical information and tear samples from patients with dry eye syndrome.
- Non-Dry eye patients (Other): Collect clinical information and tear samples from patients without dry eye syndrome.
  Interventions: Other: with/without dry eye syndrome

INTERVENTIONS:
Other: with/without dry eye syndrome — compare tear ferning structure between dry eye and non-dry eye patients
  Arms: Non-Dry eye patients

SUMMARY:
Application of tear ferning test for clinical dry eye diagnosis

DETAILED DESCRIPTION:
Comparing dry eye patients' tear ferning structure with non-dry eye patients' to develop a protocol for easy and costless diagnosis in ophthalmology.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 65 years
* For dry eye disease group:
* Schirmer's test results between 5 - 10 mm
* Tear Film Break Up Time less than 10 seconds
* Ocular Surface Disease Index of more than 25

Exclusion Criteria:

* Those have diabetes, hypertension or other chronic diseases
* No evident ocular diseases such as cornea disease, cataracts, vitreous degeneration, glaucoma, and retinopathy.
* Belong to vulnerable groups(pregnancy woman, prisoner, ethical minorities, economic or educationally disadvantaged subjects, disabled individuals such as those at terminal stage of tumorigenesis, blindness, terminal ill individuals)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Schirmer's test | 5 minutes
  to assess tear secretion volume
Tear film breakup time | 20 seconds
  to assess tear quality
Ocular surface health evaluate | 3 minutes
  To assess the health status with Lissamine green stain

SECONDARY OUTCOMES:
Ocular surface disease index | 20 minutes
  A questionnaire to assess the health status on ocular surface
  A final score is calculated which ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease.
Intraocular pressure | 2 minutes
  to determine the effects of intervention on intraocular pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Jen-Ai Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No